CLINICAL TRIAL: NCT02433262
Title: World Health Organisation (WHO) Versus International Association of Diabetes and Pregnancy Study Group (IADPSG) Diagnostic Criteria of Gestational Diabetes Mellitus and Their Associated Maternal and Neonatal Outcomes
Brief Title: WHO Versus IADPSG Diagnostic Criteria of Gestational Diabetes Mellitus and Their Associated Maternal and Neonatal Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FF-2015-067
Record Dates: First submitted 2015-04-06; First posted 2015-05-04 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — World Health Organization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WHO (World Health Organisation) (Placebo Comparator): Participants will undergo oral glucose tolerance test involving drinking of 75g glucose and blood taking for fasting and 2 hours post glucose intake. Diagnosis of GDM will be made based on these criteria:
  Fasting glucose >6 2 hour glucose >7.7
  Interventions: Other: WHO (World Health Organisation)
- IADPSG (Active Comparator): Participants will undergo oral glucose tolerance test involving drinking of 75g glucose and blood taking for fasting and 2 hours post glucose intake. Diagnosis of GDM will be made based on these criteria: (International Association of Diabetes & Pregnancy Study Group) Fasting glucose >5 2 hour glucose >8.4
  Interventions: Other: IADPSG

INTERVENTIONS:
Other: WHO (World Health Organisation) — Participants will need to undergo oral glucose tolerance test which involve drinking a 75g oral glucose. Venous blood for fasting and 2 hours post glucose intake will be taken. Diagnosis of gestational diabetes mellitus (GDM) will be made using WHO criteria. Once GDM is diagnosed, they will undergo blood sugar profile monitoring and treatment which includes diet control and/or insulin treatment if required
  Other Names: Diet control
  Arms: WHO (World Health Organisation)
Other: IADPSG — Participants will need to undergo oral glucose tolerance test which involve drinking a 75g oral glucose. Venous blood for fasting and 2 hours post glucose intake will be taken. Diagnosis of gestational diabetes mellitus (GDM) will be made using IADPSG criteria. Once GDM is diagnosed, they will undergo blood sugar profile monitoring and treatment which includes diet control and/or insulin treatment if required
  Other Names: Diet control
  Arms: IADPSG

SUMMARY:
Aim for this study is to measure the prevalence of Gestational Diabetes Mellitus (GDM) using World Health Organisation (WHO) versus International Association of Diabetes in Pregnancy Study Group (IADPSG) criteria among pregnant mother in Universiti Kebangsaan Malaysia Medical Centre (UKMMC)

DETAILED DESCRIPTION:
It will then be used to measure the incidence of adverse maternal and neonatal outcomes in women diagnosed with GDM using either of the criteria.

Patients with risk factors for GDM will be recruited and randomised to either group once fulfilled the inclusion and exclusion criteria and agreed to join this study. Subjects will then undergo 75g oral glucose tolerance test and diagnosis will be established based on the group assigned.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian citizen and able to speak and understand Malay or English
* Pregnant women with one or more risk factors for GDM between 14-37 gestational weeks
* Singleton pregnancy

Exclusion Criteria:

* Inability to complete OGTT
* Women previously diagnosed with Type 2 and Type 1 DM
* Pregnant women who refuse to participate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 506 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
To measure the prevalence of GDM diagnosed using WHO versus IADPSG criteria | 14-37weeks
  Prevalence of GDM will be reported in percentage for both groups- WHO and IADPSG

SECONDARY OUTCOMES:
To measure the incidence of adverse maternal outcomes in women diagnosed with GDM using either of the criteria (WHO or IADPSG) | 14-37 weeks
  Number of incidence in each group will be reported in percentage:
  Primary caesarean section
To measure the incidence of adverse maternal outcomes in women diagnosed with GDM using either of the criteria (WHO or IADPSG) | 14-37 weeks
  Number of incidence in each group will be reported in percentage:
  Gestational hypertension or pre-eclampsia
To measure the incidence of adverse maternal outcomes in women diagnosed with GDM using either of the criteria (WHO or IADPSG) | 14-37 weeks
  Number of incidence in each group will be reported in percentage:
  Preterm delivery (<37 weeks gestation)
To measure the incidence of adverse neonatal outcomes in women diagnosed with GDM using either of the criteria (WHO or IADPSG) | 14-37 weeks
  Number of incidence will be reported in percentage:
  Macrosomia (BW>90th centile for gestational age, gender and ethnicity)
To measure the incidence of adverse neonatal outcomes in women diagnosed with GDM using either of the criteria (WHO or IADPSG) | 14-37 weeks
  Number of incidence will be reported in percentage:
  Neonatal hypoglycaemia
To measure the incidence of adverse neonatal outcomes in women diagnosed with GDM using either of the criteria (WHO or IADPSG) | 14-37 weeks
  Number of incidence will be reported in percentage:
  Shoulder dystocia or birth injury

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics & Gynaecology Department, National University of Malaysia, Cheras, Kuala Lumpur, Malaysia